CLINICAL TRIAL: NCT05257265
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Determine the Efficacy and Safety of Once Daily Centanafadine Capsules for the Treatment of Adolescents With Attention-deficit/Hyperactivity Disorder
Brief Title: A Trial of Centanafadine Efficacy and Safety in Adolescents With Attention- Deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 405-201-00016
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: Centanafadine; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Centanafadine 164.4 mg (Experimental): Participants received centanafadine hydrochloride 164.4 milligrams (mg) XR capsules, orally, QD up to 6 weeks.
  Interventions: Drug: Centanafadine Hydrochloride
- Centanafadine 328.8 mg (Experimental): Participants received centanafadine hydrochloride 328.8 mg XR capsules, orally, QD up to 6 weeks.
  Interventions: Drug: Centanafadine Hydrochloride
- Placebo (Placebo Comparator): Participants received centanafadine matching placebo capsules, orally, QD up to 6 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Centanafadine Hydrochloride — Capsule
  Other Names: Centanafadine QD XR
  Arms: Centanafadine 164.4 mg; Centanafadine 328.8 mg
Other: Placebo — Capsule
  Other Names: Matching Placebo
  Arms: Placebo

SUMMARY:
This trial was conducted to evaluate the efficacy and safety of the Centanafadine once daily (QD) extended release (XR) capsules in adolescent participants (13 - 17 years, inclusive) with attention-deficit/hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
The trial consisted of a screening period of up to 28 days (4 weeks), a 42-day (6-week) double-blind treatment period, and a 7 (+ 2)-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 13 to 17 years (inclusive) at the time of informed consent/assent.
* A primary diagnosis of ADHD based on Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) diagnosis criteria as confirmed with the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).
* A minimum symptoms total raw score of ≥ 28 on the Attention-Deficit/Hyperactivity Disorder Rating Scale Version 5 (ADHD-RS-5) at baseline for all participants.
* A score of 4 or higher on the Clinical Global Impression - Severity - Attention Deficit/Hyperactivity Disorder (CGI-S-ADHD) at baseline.

Exclusion Criteria:

* A comorbid diagnosis of: Tourette's Disorder, Generalized Anxiety Disorder severe enough to interfere with trial procedures, Panic Disorder, Conduct Disorder, Psychosis, Post-traumatic Stress Disorder, Bipolar Disorder, Autism Spectrum Disorder, Binge Eating Disorder, Anorexia, Bulimia, Oppositional Defiant Disorder severe enough to interfere with trial conduct (allowed if it is not the primary focus of treatment), Obsessive-Compulsive Disorder severe enough to interfere with trial conduct (allowed if it is not the primary focus of treatment), or major depressive disorder (MDD) with current major depressive episode.
* Participants who are breast-feeding and/or have a positive pregnancy test result prior to receiving investigational medicinal product (IMP).
* A significant risk of committing suicide based on history and the investigator's clinical judgment, or routine psychiatric status examination, Current suicidal behavior, Imminent risk of injury to self, Active suicidal ideation. History of suicidal behavior (over the last 6 months).
* Body mass index (BMI) ≥ 40 kg/m2 or ≤ 5th percentile for age and gender based on United States (US) Centers for Disease Control and Prevention (CDC) criteria.
* Has initiated, changed, or discontinued receiving psychological interventions for ADHD within the 30 days before the screening visit, or is anticipated to start new treatment during the trial.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 459 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Attention-Deficit/Hyperactivity Disorder Rating Scale Version 5 (ADHD-RS-5) | From baseline to week 6
  Change from baseline in the ADHD-RS-5 symptoms total raw score (investigator interview with informant) at Week 6.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity - Attention-Deficit/Hyperactivity Disorder (CGI-S-ADHD) | From baseline to week 6
  Change from baseline in CGI-S-ADHD at Week 6
Conners-3 Parent Short- Change from baseline in Conners-3 Parent Short at Week 6 | From baseline to week 6

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites, contact 844-687-8522, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Ward CL, Childress AC, Jin N, Turkoglu O, Skubiak T, Wilens TE. Centanafadine for Attention-Deficit/Hyperactivity Disorder in Adolescents: A Randomized Clinical Trial. J Am Acad Child Adolesc Psychiatry. 2025 Jul 4:S0890-8567(25)00327-2. doi: 10.1016/j.jaac.2025.06.023. Online ahead of print. PMID 40619095